CLINICAL TRIAL: NCT04703712
Title: Effectiveness of Lens Extraction Combined With Goniosynechialysis Versus Trabeculectomy in Treating Advanced Angle-closure Glaucoma: a Randomized Controlled Trial
Brief Title: Lens Extraction Combined With Goniosynechialysis Versus Trabeculectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Yuhong Chen, Professor, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAC Glaucoma
Record Dates: First submitted 2021-01-03; First posted 2021-01-11 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Glaucoma, Angle-Closure
Keywords: phacoemulsification; goniosynechialysis; trabeculectomy
MeSH Terms: conditions — Glaucoma, Angle-Closure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lens extraction combined with goniosynechialysis group (Active Comparator): One hundred and fifty-eight patients with advanced angle-closure glaucoma underwent phacoemulsification combined with goniosynechialysis.
  Interventions: Procedure: Lens extraction combined with goniosynechialysis
- Trabeculectomy Group (Active Comparator): One hundred and fifty-eight patients with advanced angle-closure glaucoma underwent trabeculectomy.
  Interventions: Procedure: Trabeculectomy surgery

INTERVENTIONS:
Procedure: Lens extraction combined with goniosynechialysis — The patients enrolled underwent phacoemulsification combined with goniosynechialysis surgery.
  Arms: Lens extraction combined with goniosynechialysis group
Procedure: Trabeculectomy surgery — The patients enrolled underwent trabeculectomy surgery
  Arms: Trabeculectomy Group

SUMMARY:
To compare the effectiveness of lens extraction combined with goniosynechialysis and trabeculectomy in treating advanced angle-closure glaucoma.

DETAILED DESCRIPTION:
Advanced angle closure glaucoma (AACG) can result in severe visual function defect or even blindness with or without acute attacks. Different from open angle glaucoma (OAG), the main principle of treatment for AACG is not only to lower intraocular pressure (IOP) but also to protect the anterior chamber angle from closing. Previously, the most common and classical treatment for AACG was trabeculectomy. However, both doctors and patients are not satisfied with this surgery because of its limited success rate due to fibrosis of the filtration pathway. Besides, trabeculectomy has various complications, such as shallow anterior chamber, choroidal effusion, suprachoroidal hemorrhage, malignant glaucoma, and bleb leakage associated endophthalmitis. In addition, patients who underwent trabeculectomy will have decreased visual acuity in a couple of years due to accelerated development of cataract. Since a thickened and anterior-positioned lens could play a crucial role in the pathogenesis of AACG, cataract surgery has also been used. Accumulative evidence shows lens extraction alone is an efficient way in treating the early stage of ACG but has limited success rate in AACG. Lens extraction combined with goniosynechialysis (LEG) has been proved to be better than lens extraction alone in re-opening the anterior chamber angle for ACG patients with extensive peripheral anterior synechia and possibly have better effect than trabeculectomy as well from our preliminary data, which has not been proved yet. Thus, this investigation is designed to compare the effect of LEG and trabeculectomy in AACG patients prospectively in 3 years of follow-up. The investigators hypothesize that LEG could have better IOP control and better visual function than trabeculectomy in long term for AACG patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 years old to 80 years old
2. more than 180-degree synechial closure of anterior chamber angle on gonioscopy
3. IOP higher than 21mmHg under the use of more than two anti-glaucoma eye drops
4. mean deviation of visual field worse than -12dB on Humphrey 24-2
5. phakic eyes

Exclusion Criteria:

1. Snellen visual acuity worse than 0.02
2. history of ocular trauma
3. uveitis
4. previous ocular surgeries
5. significant conjunctival scar
6. visible neovascular on iris or anterior chamber angle
7. other severe eye diseases that would affect visual function significantly, such as age-related macular degeneration and pathogenic myopia.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2021-01-30 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) change at one month | one month
  Change from baseline IOP after phacoemulsification combined with goniosynechialysis or trabeculectomy at one month.
IOP change at three months | three months
  Change from baseline IOP after phacoemulsification combined with goniosynechialysis or trabeculectomy at three months.
IOP change at six months | six months
  Change from baseline IOP after phacoemulsification combined with goniosynechialysis or trabeculectomy at six months.
IOP change at one year | one year
  Change from baseline IOP after phacoemulsification combined with goniosynechialysis or trabeculectomy at one year.
IOP change at two years | two years
  Change from baseline IOP after phacoemulsification combined with goniosynechialysis or trabeculectomy at two years.
IOP change at three years | three years
  Change from baseline IOP after phacoemulsification combined with goniosynechialysis or trabeculectomy at three years.
Best corrected visual acuity at one month | one month
  Best corrected visual acuity of participants after surgery at one month
Best corrected visual acuity at three months | three months
  Best corrected visual acuity of participants after surgery at three months
Best corrected visual acuity at six months | six months
  Best corrected visual acuity of participants after surgery at six months
Best corrected visual acuity at one year | one year
  Best corrected visual acuity of participants after surgery at one year
Best corrected visual acuity at two years | two years
  Best corrected visual acuity of participants after surgery at two years
Best corrected visual acuity at three years | three years
  Best corrected visual acuity of participants after surgery at three years

SECONDARY OUTCOMES:
Mean deviation | one month, three months, six months, one year, two years, three years
  The mean deviation value of Humphery visual filed tests before and after surgery.
The thickness of retinal nerve fiber layer (RNFL) | one month, three months, six months, one year, two years, three years
  The RNFL thickness measured by optical coherence topography (OCT)
The thickness of ganglion cell complex (GCC) | one month, three months, six months, one year, two years, three years
  The GCC thickness measured by OCT
Number of eye drops | one month, three months, six months, one year, two years, three years
  The number of eye drops after surgery.
Adverse event | one month, three months, six months, one year, two years, three years
  Adverse events of each group, such as cornea edma, ocular hypotension, hemorrhage

CONTACTS AND LOCATIONS:
Locations (1):
- Eye & ENT Hospital, Shanghai, China